CLINICAL TRIAL: NCT01473966
Title: Coffee Against Obstipation in Intensive Care Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Christoph Eisenbach, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COFFEE
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Obstipation
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard of care (No Intervention): patients receive standard care
- Coffee orally (Experimental): patients will receive standard of care plus coffee orally
  Interventions: Dietary Supplement: coffee
- coffee rectally (Experimental): patients receive standard of care plus coffee rectally
  Interventions: Dietary Supplement: coffee rectally

INTERVENTIONS:
Dietary Supplement: coffee — patients will receive a cup of coffee at room temperature orally twice daily
  Arms: Coffee orally
Dietary Supplement: coffee rectally — patients receive an enema of two cups of coffee at room temperature once daily
  Other Names: Coffee
  Arms: coffee rectally

SUMMARY:
Coffee might stimulate bowel movement and thus overcome obstipation in intensive care unit (ICU) patients.

DETAILED DESCRIPTION:
Critically ill patients requiring ventilator support frequently suffer from obstipation. We hypothesize that coffee, administered either orally or rectally, might stimulate bowel movement.

ELIGIBILITY:
Inclusion Criteria:

* admission to the medical intensive care unit of the Dept. of Gastroenterology at the university hospital heidelberg
* requires ventilator support for an anticipated more than 72 hours
* age older than 18 years

Exclusion Criteria:

* pregnancy
* known allergy to coffee
* mechanical ileus
* presence of enterostoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Bowel movement rate | participants will be followed for the duration of hospital stay, an expected average of 5 weeks

SECONDARY OUTCOMES:
time on mechanical ventilation | participants will be followed for the duration of intensive care unit stay, an expected average of 3 weeks
time of stay on ICU | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
lengths of hospitalisation | an average of 5 weeks of hospital stay is expected
in hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
long term mortality | 6 months following discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Eisenbach, Principal Investigator — University of Heidelberg, Heidelberg, Germany
Locations (1):
- University hospital of Heidelberg, Heidelberg, Germany